CLINICAL TRIAL: NCT03489317
Title: Gut Microbiomes and Viromes in Patients With Metabolic Syndrome
Brief Title: Gut Microbiomes in Patients With Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yeoh Yun Kit, Research Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2017.514
Record Dates: First submitted 2018-03-23; First posted 2018-04-05 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Syndrome
Keywords: gut microbiome; stool
MeSH Terms: conditions — Metabolic Syndrome | interventions — Metformin; Simvastatin; Amlodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stools, whole blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No metabolic syndrome: Participants who do not fulfill any of the five criteria for metabolic syndrome defined by the International Diabetes Federation.
- Metabolic syndrome- partial: Participants who fulfill one or two of the five criteria for metabolic syndrome defined by the International Diabetes Federation.
  Interventions: Drug: Metformin; Behavioral: lifestyle modification; Drug: Simvastatin 10mg; Drug: Amlodipine 5mg
- Metabolic syndrome- full: Participants who fulfill three or more of the five criteria for metabolic syndrome defined by the International Diabetes Federation.
  Interventions: Drug: Metformin; Behavioral: lifestyle modification; Drug: Simvastatin 10mg; Drug: Amlodipine 5mg

INTERVENTIONS:
Drug: Metformin — Participants with high glucose levels will usually be prescribed Metformin 250 mg three times daily. Can be prescribed to either metabolic syndrome-partial or full groups depending on their metabolic syndrome conditions.
  Groups: Metabolic syndrome- full; Metabolic syndrome- partial
Behavioral: lifestyle modification — Participants with metabolic syndrome will be offered advice on modifying their diets and exercise regimes. Can be prescribed to either metabolic syndrome-partial or full groups depending on their metabolic syndrome conditions.
  Groups: Metabolic syndrome- full; Metabolic syndrome- partial
Drug: Simvastatin 10mg — Participants with elevated lipid levels will usually be prescribed simvastatin 10 mg at night. Can be prescribed to either metabolic syndrome-partial or full groups depending on their metabolic syndrome conditions.
  Groups: Metabolic syndrome- full; Metabolic syndrome- partial
Drug: Amlodipine 5mg — Participants with high blood pressure could be prescribed antihypertensive medicine such as Amlodipine. Can be prescribed to either metabolic syndrome-partial or full groups depending on their metabolic syndrome conditions.
  Groups: Metabolic syndrome- full; Metabolic syndrome- partial

SUMMARY:
Metabolic syndrome (MS) is defined by a manifestation of cardiometabolic risk factors including high blood pressure, glucose and triglycerides, low high-density lipoprotein (HDL) cholesterol, and abdominal obesity. It is closely associated with other diseases such as fatty liver and gouty arthritis. In recent years there is evidence that gut microorganisms are intimately linked to health and wellbeing. Here, the investigators hypothesize that gut microorganisms are involved in the regulation and/or onset of MS and its symptoms.

DETAILED DESCRIPTION:
There is mounting evidence that the gut microbiome plays a vital role in health and wellbeing. In particular, population-association and mouse model studies have demonstrated that gut bacteria can be reproducibly linked to obesity and diabetes. There is, however, a lack of progress in translating current scientific knowledge to healthcare practices in part due to the strong influence of biogeography and demography on gut microbiomes. Another major knowledge gap in gut microbiomes is the ecology of gut viruses and their associations with MS despite having intimate relationships with human and bacterial hosts.

In this study, the investigators aim to assess variation in the gut microbiomes of patients with MS with reference to the healthy population in Hong Kong, and to explore gut microorganisms as predictive/diagnostic markers of MS and clinical outcomes associated with medical interventions. This will be achieved through studying microorganisms in the stools of participants. The investigators will use the 16S small subunit ribosomal RNA (16S rRNA) marker gene to create compositional profiles of the gut microbial community in healthy and individuals with MS to identify bacterial populations that are associated with the onset and progression of MS. A subset of samples will be selected for bulk DNA sequencing based on their stool community profiles and/or MS parameters to obtain genomic information of the microorganisms involved.

Participants who undergo intervention as part of their routine medical care for MS will be invited to provide stool samples following intervention. These stools will be used to profile gut microbial communities to investigate whether their compositions undergo changes reflective of medical intervention. Here, the aim is to investigate whether resolution of MS symptoms can be linked to alterations in gut microorganisms, and the hypothesis is that their profiles will more closely resemble healthy individuals following medical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Hong Kong

Exclusion Criteria:

* Major organ system impairment such as heart failure, renal failure, and severe impairment of respiratory function.
* On long-term regular immunosuppressive therapy
* Current or history of malignancy
* Current or history of major gastrointestinal diseases, including inflammatory bowel disease, major gastrointestinal surgery
* On medication for glucose or lipid control, such as metformin and statin

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Hong Kong will be invited from health talks, blogs, notices and advertisement through various public media channels, as well as patients referred to the Lek Yuen Health Centre, a university teaching clinic, for suspected or confirmed metabolic syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in waist circumference at four weeks | four weeks in participants receiving drug intervention for metabolic syndrome
  Waist circumference is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a circumference of ≥90 cm (male) or ≥80 cm (female) is a criteria for metabolic syndrome. The investigators will measure this in participants receiving drug-based treatment before and four weeks after medical intervention, and assess stool microbial community compositions to determine whether any changes in waist circumference can be associated with gut microorganisms.
Change in baseline systolic and diastolic blood pressure at four weeks | four weeks in participants receiving drug intervention for metabolic syndrome
  Blood pressure is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a blood pressure reading of ≥130/85 mm Hg (systolic/diastolic pressure) is a criteria for metabolic syndrome. The investigators will measure this in participants receiving drug-based treatment before and four weeks after medical intervention, and assess stool microbial community compositions to determine whether any changes in baseline systolic and diastolic blood pressure can be associated with gut microorganisms.
Change in blood triglyceride levels at four weeks | four weeks in participants receiving drug intervention for metabolic syndrome
  Blood triglyceride concentration is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a triglyceride level of ≥1.7 mmol/L is a criteria for metabolic syndrome. The investigators will measure this in participants receiving drug-based treatment before and four weeks after medical intervention, and assess stool microbial community compositions to determine whether any changes in blood triglyceride levels can be associated with gut microorganisms.
Change in high-density lipoprotein (HDL) cholesterol levels at four weeks | four weeks in participants receiving drug intervention for metabolic syndrome
  High-density lipoprotein (HDL) cholesterol levels is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a HDL cholesterol level of <1.03 mmol/L (males) or <1.29 mmol/L (females) is a criteria for metabolic syndrome. The investigators will measure this in participants receiving drug-based treatment before and four weeks after medical intervention, and assess stool microbial community compositions to determine whether HDL cholesterol levels can be associated with gut microorganisms.
Change in fasting blood sugar levels at four weeks | four weeks in participants receiving drug intervention for metabolic syndrome
  Fasting blood sugar levels is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a fasting blood sugar level of ≥5.6 mmol/L is a criteria for metabolic syndrome. The investigators will measure this in participants receiving drug-based treatment before and four weeks after medical intervention, and assess stool microbial community compositions to determine whether fasting blood sugar levels can be associated with gut microorganisms.
Change in waist circumference at six months | six months in all participants with metabolic syndrome
  Waist circumference is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a circumference of ≥90 cm (male) or ≥80 cm (female) is a criteria for metabolic syndrome. The investigators will measure this in all participants with metabolic syndrome six months after their initial visit, and assess stool microbial community compositions to determine whether any changes in waist circumference can be associated with gut microorganisms.
Change in baseline systolic and diastolic blood pressure at six months | six months in all participants with metabolic syndrome
  Blood pressure is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a blood pressure reading of ≥130/85 mm Hg (systolic/diastolic pressure) is a criteria for metabolic syndrome. The investigators will measure this in all participants with metabolic syndrome six months after their initial visit, and assess stool microbial community compositions to determine whether any changes in baseline systolic and diastolic blood pressure can be associated with gut microorganisms.
Change in blood triglyceride levels at six months | six months in all participants with metabolic syndrome
  Blood triglyceride concentration is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a triglyceride level of ≥1.7 mmol/L is a criteria for metabolic syndrome. The investigators will measure this in all participants with metabolic syndrome six months after their initial visit, and assess stool microbial community compositions to determine whether any changes in blood triglyceride levels can be associated with gut microorganisms.
Change in high-density lipoprotein (HDL) cholesterol levels at six months | six months in all participants with metabolic syndrome
  High-density lipoprotein (HDL) cholesterol levels is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a HDL cholesterol level of <1.03 mmol/L (males) or <1.29 mmol/L (females) is a criteria for metabolic syndrome. The investigators will measure this in all participants with metabolic syndrome six months after their initial visit, and assess stool microbial community compositions to determine whether HDL cholesterol levels can be associated with gut microorganisms.
Change in fasting blood sugar levels at six months | six months in all participants with metabolic syndrome
  Fasting blood sugar levels is one of the five criteria for classifying metabolic syndrome as defined by the International Diabetes Federation. Specifically, a fasting blood sugar level of ≥5.6 mmol/L is a criteria for metabolic syndrome. The investigators will measure this in all participants with metabolic syndrome six months after their initial visit, and assess stool microbial community compositions to determine whether fasting blood sugar levels can be associated with gut microorganisms.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kit Yeoh, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Microbiology, Chinese University of Hong Kong, Shatin
  - Lek Yuen Health Centre, Shatin

IPD SHARING:
Plan to Share IPD: Undecided
Participant data may be shared with researchers within the Faculty of Medicine at the Chinese University of Hong Kong, however, these will likely be limited to the healthy cohort as controls for other gut community surveys or the metabolic syndrome cohort for research into closely related medical conditions such as hypertension.
  The investigators will share participant clinical (blood pressure, waist circumference, fasting blood sugar, triglycerides), demography (age, gender, medical history, etc) and gut microbial community composition data within the department where the need arises and appropriate approvals have been obtained.

DOCUMENTS (1):
  • Study Protocol (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03489317/Prot_000.pdf